CLINICAL TRIAL: NCT00760877
Title: An Open Label, Randomized Study of Nilotinib vs. Standard Imatinib (400/600 mg QD) Comparing the Kinetics of Complete Molecular Response for CML-CP Patients With Evidence of Persistent Leukemia by RQ-PCR.
Brief Title: Nilotinib Versus Standard Imatinib (400/600 mg Every Day (QD)) Comparing the Kinetics of Complete Molecular Response for Chronic Myelogenous Leukemia in Chronic Phase (CML-CP) Pts With Evidence of Persistent Leukemia by Real-time Quantitative Polymerase Chain Reaction (RQ-PCR)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAMN107A2405; 2009-012616-40 (EudraCT Number)
Record Dates: First submitted 2008-09-25; First posted 2008-09-26 (Estimated); Results first posted 2016-08-16 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-10

CONDITIONS: CHRONIC MYELOGENOUS LEUKEMIA
Keywords: MYELOGENOUS; LEUKEMIA; Chronic Phase; CML
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia | interventions — nilotinib; Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nilotinib (Experimental): Participants received Nilotinib 400 mg orally twice daily (bid) for 48 months.
  Interventions: Drug: Nilotinib
- Imatinib (Active Comparator): Participants received Imatinib 400 mg or 600 mg once daily (qd) (based on the participant's dose prior to randomization) for 48 months.
  Interventions: Drug: Imatinib

INTERVENTIONS:
Drug: Nilotinib — Supplied in 200 mg capsules
  Arms: Nilotinib
Drug: Imatinib — Supplied in 100 mg and 400 mg capsules
  Other Names: Glivec/Gleevec
  Arms: Imatinib

SUMMARY:
The primary goal of this study was to determine the rate of confirmed best cumulative complete molecular response (CMR) within the first year of study therapy with imatinib or nilotinib. The study also explored the impact and significance of the achieved CMR on patient outcomes (progression free survival (PFS), event free survival (EFS) and overall survival (OS), characterized the kinetics of CMR achieved in both treatment arms and after the cross-over.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of chronic myeloid leukemia associated with BCR-ABL quantifiable by RQ-PCR Documented CCyR by bone marrow or BCR-ABL<1% IS in the past 12 months Persistent disease demonstrated by two PCR positive tests 3 months apart both during the past 6 months.

Treatment with imatinib for at least 2 years with 400 mg or 600 mg and a stable dose No other current or planned anti-leukemia therapies

Exclusion Criteria:

Patient has evidence of rising PCR (a confirmed >1 log increase in previous 6 months) Patient has received another investigational agent within last 6 months or tyrosine kinase inhibitors (TKIs) other than imatinib Prior allogeneic stem cell transplantation

Impaired cardiac function including any one of the following:

Inability to monitor the QT interval on electrocardiogram (ECG) Long QT syndrome or a known family history of long QT syndrome. Clinically significant resting brachycardia (<50 beats per minute) QTc > 450 msec on baseline ECG (using the QTcF formula). If QTcF >450 msec and electrolytes are not within normal ranges, electrolytes should be corrected and then the patient re-screened for QTc Myocardial infarction within 12 months prior to starting study Other clinically significant uncontrolled heart disease (e.g. unstable angina, congestive heart failure or uncontrolled hypertension) History of or presence of clinically significant ventricular or atrial tachyarrhythmias Administration of cytokine therapy (e.g. G-CSF, GM-CSF or SCF) within 4 weeks prior to study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2009-06; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (29):
- Novartis Investigative Site, Caba, Buenos Aires, Argentina
- Australia (9):
  - Novartis Investigative Site, St Leonards, New South Wales
  - Novartis Investigative Site, Westmead, New South Wales
  - Novartis Investigative Site, Herston, Queensland
  - Novartis Investigative Site, South Brisbane, Queensland
  - Novartis Investigative Site, Woolloongabba, Queensland
  - Novartis Investigative Site, Adelaide, South Australia
  - Novartis Investigative Site, Parkville, Victoria
  - Novartis Investigative Site, Prahran, Victoria
  - Novartis Investigative Site, Nedlands, Western Australia
- Brazil (5):
  - Novartis Investigative Site, Belo Horizonte, Minas Gerais
  - Novartis Investigative Site, Curitiba, Paraná
  - Novartis Investigative Site, Rio de Janeiro, Rio de Janeiro
  - Novartis Investigative Site, Campinas, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
- Canada (5):
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Hamilton, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Québec, Quebec
- France (5):
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Créteil
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Vandœuvre-lès-Nancy
- Spain (4):
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Madrid, Madrid
  - Novartis Investigative Site, Pamplona, Navarre

REFERENCES:
- [Derived] Hughes TP, Lipton JH, Spector N, Cervantes F, Pasquini R, Clementino NC, Dorlhiac Llacer PE, Schwarer AP, Mahon FX, Rea D, Branford S, Purkayastha D, Collins L, Szczudlo T, Leber B. Deep molecular responses achieved in patients with CML-CP who are switched to nilotinib after long-term imatinib. Blood. 2014 Jul 31;124(5):729-36. doi: 10.1182/blood-2013-12-544015. Epub 2014 Jun 19. PMID 24948656

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomized 1:1. Participants in the imatinib arm were permitted to cross-over to nilotinib after 2 years on study if complete molecular response (CMR) was not achieved, or at any time during the study if participants experienced treatment failure, had confirmed loss of major molecular response (MMR) or had confirmed loss of CMR.
Period: Overall Study
Arm/Group | Nilotinib | Imatinib
Started | 104 | 103
Cross-over to Nilotinib | 0 (Not applicable: cross-over occurred from imatinib to nilotinib only.) | 46
Safety Set | 101 | 103
Completed | 59 | 77
Not Completed | 45 | 26
Not completed — Protocol Violation | 1 | 0
Not completed — Non-compliance with protocol treatment | 2 | 1
Not completed — Pregnancy | 1 | 4
Not completed — Death | 2 | 1
Not completed — Withdrawal by Subject | 7 | 3
Not completed — Adverse Event | 19 | 12
Not completed — Participant diagnosed with AML | 0 | 1
Not completed — Participant not eligible to cross-over | 0 | 1
Not completed — Physician Decision | 1 | 2
Not completed — Participants transferred to AMN107A2408 | 11 | 1
Not completed — Treatment failure | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nilotinib | Imatinib | Total
Number analyzed (Participants) | 104 | 103 | 207
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.3 (13.26) | 49.9 (13.07) | 49.1 (13.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 38 | 71
  Male | 71 | 65 | 136

OUTCOME MEASURES:

1. Primary Outcome: Rate of Confirmed Best Cumulative Complete Molecular Response (CMR)
Description: The rate of confirmed best cumulative CMR was defined as the number of participants who had confirmed CMR during the first 12 months of treatment after the randomization date. Participants who achieved confirmed best cumulative CMR during the first 12 months were considered responders. Participants who dropped out early or who did not provide sufficient data for any reason were considered to be non-responders. The definition of CMR is undetectable BCR-ABL (fusion gene formed between bcr gene from chromosome 22 and abl gene from chromosome 9) where BCR-ABL ratio in % international scale (IS) ≤ 0.00001 by real-time quantitative polymerase chain reaction (RQ-PCR) where there was no detectable BCR-ABL and 1) the test had a sensitivity of at least 4.5 logs below the standardized baseline; 2) RQ-PCR negativity was confirmed on the next RQ-PCR sample (usually 3 months later); and 3) the date of confirmed CMR was the date of the first of two negative results with sensitivity >4.5 logs.
Time Frame: 12 months
Population: The intent-to-treat analysis set, which included all randomized participants, was analyzed.
Measure: Number; unit: Participants
Arm/Group | Nilotinib | Imatinib
Number analyzed (Participants) | 104 | 103
Participants
  Responders | 13 | 6
  Non-responders | 91 | 97
Statistical Analysis 1: Comparison: Nilotinib vs Imatinib; Test type: Superiority or Other; p = 0.1083, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 2.096, 95% CI 2-sided [0.766 to 5.738]

2. Secondary Outcome: Rate of Confirmed Best Cumulative CMR
Description: The rate of confirmed best cumulative CMR was defined as the number of participants who had confirmed CMR during the 24, 36 and 48 months post treatment after the randomization date. Participants who achieved confirmed best cumulative CMR during the first 12 months were considered responders. Participants who dropped out early or who did not provide sufficient data for any reason were considered to be non-responders. The definition of CMR is undetectable BCR-ABL (fusion gene formed between bcr gene from chromosome 22 and abl gene from chromosome 9) where BCR-ABL ratio in % international scale (IS) ≤ 0.00001 by RQ-PCR where there was no detectable BCR-ABL and 1) the test had a sensitivity of at least 4.5 logs below the standardized baseline; 2) RQ-PCR negativity was confirmed on the next RQ-PCR sample (usually 3 months later); and 3) the date of confirmed CMR was the date of the first of two negative results with sensitivity >4.5 logs.
Time Frame: 24 months, 36 month, 48 months
Population: The intent-to-treat analysis set, which included all randomized participants, was analyzed.
Measure: Number; unit: Participants
Arm/Group | Nilotinib | Imatinib
Number analyzed (Participants) | 104 | 103
Participants
  24 months, Responders | 24 | 11
  24 months, Non-responders | 80 | 92
  36 months, Responders | 29 | 21
  36 months, Non-responders | 75 | 82
  48 months, Responders | 32 | 21
  48 months, Non-responders | 72 | 82

3. Secondary Outcome: Number of Cross-over Participants With CMR
Description: The definition of CMR is undetectable BCR-ABL (fusion gene formed between bcr gene from chromosome 22 and abl gene from chromosome 9) where BCR-ABL ratio in % international scale (IS) ≤ 0.00001 by RQ-PCR where there was no detectable BCR-ABL and 1) the test had a sensitivity of at least 4.5 logs below the standardized baseline; 2) RQ-PCR negativity was confirmed on the next RQ-PCR sample (usually 3 months later); and 3) the date of confirmed CMR was the date of the first of two negative results with sensitivity >4.5 logs.
Time Frame: 24 months, 36 months, 48 months
Population: Participants from the Imatinib treatment group who crossed over to the Nilotinib treatment group were analyzed.
Measure: Number; unit: Participants
Arm/Group | Nilotinib
Number analyzed (Participants) | 46
Participants
  24 months | 3
  36 months | 6
  48 months | 9

4. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time from the date of randomization to the date of the earliest documented progression-defining event as follows: transformation to blast crisis or accelerated phase disease, or death from any cause.
Time Frame: 48 months
Population: 24 months, Non-responders
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nilotinib | Imatinib
Number analyzed (Participants) | 104 | 103
months | NA [NA to NA] — The median and 95% confidence interval (CI) could not be calculated because there were too few events. | NA [NA to NA] — The median and 95% CI could not be calculated because there were too few events.

5. Secondary Outcome: Event-free Survival
Description: Event-free survival was defined as the time from the date of randomization to the date of first occurrence of any of the following events on study treatment: loss of complete hematological response, confirmed loss of complete cytogenetic response (CCyR), confirmed loss of major molecular response (MMR), death from any cause during treatment, progression to the accelerated phase or blast crisis of chronic myelogenous leukemia (CML) per European Leukemia Network (ELN) criteria, whichever was earliest.
Time Frame: 48 months
Population: The intent-to-treat analysis set, which included all randomized participants, was analyzed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nilotinib | Imatinib
Number analyzed (Participants) | 104 | 103
Months | NA [NA to NA] — The median and 95% CI could not be calculated because there were too few events. | NA [NA to NA] — The median and 95% CI could not be calculated because there were too few events.

6. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time from the date of randomization to the date of death due to any cause at any time during the study, including the follow-up period after discontinuation of treatment.
Time Frame: 48 months
Population: The intent-to-treat analysis set, which included all randomized participants, was analyzed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nilotinib | Imatinib
Number analyzed (Participants) | 104 | 103
Months | NA [NA to NA] — The median and 95% CI could not be calculated because there were too few events. | NA [NA to NA] — The median and 95% CI could not be calculated because there were too few events.

ADVERSE EVENTS:
Groups:
- Nilotinib: Nilotinib
- Imatinib: Imatinib
- Imatinib Subset That Crossed Over to Nilotinib: Imatinib subset that crossed over to nilotinib
Arm/Group | Nilotinib | Imatinib | Imatinib Subset That Crossed Over to Nilotinib
Serious Adverse Events (participants affected / at risk) | 21/101 | 16/103 | 8/46
Other Adverse Events (participants affected / at risk) | 99/101 | 79/103 | 39/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nilotinib (N=101) | Imatinib (N=103) | Imatinib Subset That Crossed Over to Nilotinib (N=46)
ACUTE CORONARY SYNDROME (Cardiac disorders) | 1 | 0 | 1
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1 | 0 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 1 | 2 | 0
ATRIAL FLUTTER (Cardiac disorders) | 0 | 0 | 1
CARDIOPULMONARY FAILURE (Cardiac disorders) | 1 | 0 | 0
CORONARY ARTERY DISEASE (Cardiac disorders) | 1 | 0 | 0
LEFT VENTRICULAR DYSFUNCTION (Cardiac disorders) | 0 | 1 | 0
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 1 | 0
PERICARDITIS (Cardiac disorders) | 0 | 1 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 | 0 | 0
ANAL FISSURE (Gastrointestinal disorders) | 0 | 0 | 1
CROHN'S DISEASE (Gastrointestinal disorders) | 1 | 0 | 0
INGUINAL HERNIA (Gastrointestinal disorders) | 0 | 1 | 0
INFLUENZA LIKE ILLNESS (General disorders) | 1 | 0 | 0
PYREXIA (General disorders) | 0 | 0 | 1
CHOLECYSTITIS (Hepatobiliary disorders) | 0 | 0 | 1
CHOLELITHIASIS (Hepatobiliary disorders) | 1 | 1 | 0
CELLULITIS (Infections and infestations) | 0 | 2 | 0
ERYSIPELAS (Infections and infestations) | 1 | 0 | 0
INFECTED SKIN ULCER (Infections and infestations) | 1 | 0 | 0
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 0 | 0
LUNG INFECTION (Infections and infestations) | 0 | 1 | 0
OSTEOMYELITIS (Infections and infestations) | 1 | 0 | 0
PNEUMONIA (Infections and infestations) | 0 | 1 | 1
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0
BACK INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 1
DRUG ADMINISTRATION ERROR (Injury, poisoning and procedural complications) | 0 | 0 | 1
LIGAMENT RUPTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0
MUSCLE INJURY (Injury, poisoning and procedural complications) | 1 | 0 | 0
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
SPINAL COLUMN STENOSIS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
ACUTE MYELOID LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
METASTASES TO PERITONEUM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
NON-SMALL CELL LUNG CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
RENAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
CEREBRAL ARTERY OCCLUSION (Nervous system disorders) | 1 | 0 | 0
CEREBRAL ISCHAEMIA (Nervous system disorders) | 1 | 0 | 0
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 | 0 | 1
EMBOLIC STROKE (Nervous system disorders) | 1 | 0 | 0
BLADDER DILATATION (Renal and urinary disorders) | 1 | 0 | 0
NEPHROLITHIASIS (Renal and urinary disorders) | 0 | 2 | 0
URINARY RETENTION (Renal and urinary disorders) | 0 | 1 | 0
LUNG DISORDER (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 | 1 | 0
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 1 | 0 | 0
PERIPHERAL VASCULAR DISORDER (Vascular disorders) | 0 | 0 | 1
VASCULITIS (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nilotinib (N=101) | Imatinib (N=103) | Imatinib Subset That Crossed Over to Nilotinib (N=46)
ANAEMIA (Blood and lymphatic system disorders) | 6 | 12 | 5
CONJUNCTIVAL HAEMORRHAGE (Eye disorders) | 1 | 6 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 12 | 8 | 5
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 13 | 7 | 5
CONSTIPATION (Gastrointestinal disorders) | 15 | 0 | 3
DIARRHOEA (Gastrointestinal disorders) | 14 | 19 | 4
NAUSEA (Gastrointestinal disorders) | 22 | 16 | 4
VOMITING (Gastrointestinal disorders) | 11 | 6 | 0
ASTHENIA (General disorders) | 9 | 4 | 5
FATIGUE (General disorders) | 16 | 8 | 6
INFLUENZA LIKE ILLNESS (General disorders) | 7 | 3 | 2
OEDEMA PERIPHERAL (General disorders) | 6 | 7 | 1
PAIN (General disorders) | 7 | 3 | 1
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 10 | 0 | 6
FOLLICULITIS (Infections and infestations) | 8 | 0 | 2
INFLUENZA (Infections and infestations) | 9 | 9 | 2
NASOPHARYNGITIS (Infections and infestations) | 9 | 5 | 2
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 20 | 14 | 7
URINARY TRACT INFECTION (Infections and infestations) | 8 | 1 | 2
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 19 | 5 | 8
AMYLASE INCREASED (Investigations) | 9 | 7 | 2
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 14 | 10 | 6
BILIRUBIN CONJUGATED INCREASED (Investigations) | 4 | 0 | 4
BLOOD BILIRUBIN INCREASED (Investigations) | 10 | 1 | 2
BLOOD CHOLESTEROL INCREASED (Investigations) | 8 | 2 | 0
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 1 | 9 | 2
BLOOD CREATININE INCREASED (Investigations) | 6 | 10 | 2
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 8 | 2 | 2
GLOBULINS DECREASED (Investigations) | 4 | 8 | 0
HIGH DENSITY LIPOPROTEIN DECREASED (Investigations) | 2 | 6 | 3
LIPASE INCREASED (Investigations) | 19 | 13 | 7
LOW DENSITY LIPOPROTEIN INCREASED (Investigations) | 2 | 3 | 4
WEIGHT DECREASED (Investigations) | 10 | 5 | 2
DECREASED APPETITE (Metabolism and nutrition disorders) | 8 | 6 | 1
HYPERCHOLESTEROLAEMIA (Metabolism and nutrition disorders) | 11 | 6 | 7
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 4 | 6 | 6
HYPERTRIGLYCERIDAEMIA (Metabolism and nutrition disorders) | 3 | 7 | 2
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 9 | 13 | 7
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 16 | 10 | 6
BACK PAIN (Musculoskeletal and connective tissue disorders) | 12 | 9 | 7
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 15 | 18 | 1
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 10 | 8 | 2
MYALGIA (Musculoskeletal and connective tissue disorders) | 14 | 2 | 6
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 14 | 4 | 8
DIZZINESS (Nervous system disorders) | 5 | 6 | 3
HEADACHE (Nervous system disorders) | 43 | 13 | 8
DEPRESSION (Psychiatric disorders) | 6 | 4 | 2
INSOMNIA (Psychiatric disorders) | 12 | 5 | 2
COUGH (Respiratory, thoracic and mediastinal disorders) | 11 | 9 | 4
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 3
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 6 | 6 | 0
ALOPECIA (Skin and subcutaneous tissue disorders) | 11 | 0 | 4
DRY SKIN (Skin and subcutaneous tissue disorders) | 20 | 0 | 3
PRURITUS (Skin and subcutaneous tissue disorders) | 30 | 0 | 2
RASH (Skin and subcutaneous tissue disorders) | 30 | 4 | 9
RASH FOLLICULAR (Skin and subcutaneous tissue disorders) | 4 | 0 | 3
HYPERTENSION (Vascular disorders) | 10 | 6 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.